CLINICAL TRIAL: NCT06392958
Title: Application of Improved Baduanjin Combined Cross-theoretical Model Based on Internet in Family Empowering Elderly PCI Cardiac Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: KY-2024-034
Record Dates: First submitted 2024-04-11; First posted 2024-05-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-04

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; ba duan jin; Cross-theoretical model; Family empowerment
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Routine nursing: including pre-operation and 1d before discharge self-health management lectures on cardiac rehabilitation, mainly according to the essentials of China's Guidelines for Cardiac Rehabilitation and Secondary Prevention 2018, and the distribution of the knowledge manual of five major prescriptions for cardiac rehabilitation; After discharge, patients were followed up 1 month, 3 months and 6 months after surgery, including medication compliance, exercise diet, review reminder and other issues, and provided guidance on the problems existing in patients.
- Test group A (Experimental): Conventional intervention means + Internet platform improved Baduanjin intervention method
  Interventions: Other: Traditional Chinese Medicine exercises - Baduanjin
- Test group B (Experimental): Family empowering cardiac rehabilitation management under conventional intervention + cross-theoretical model
  Interventions: Other: Traditional Chinese Medicine exercises - Baduanjin
- Test group C (Experimental): Conventional intervention means + Internet platform improvement Baduanjin + cross-theoretical model of family empowerment cardiac rehabilitation management
  Interventions: Other: Traditional Chinese Medicine exercises - Baduanjin

INTERVENTIONS:
Other: Traditional Chinese Medicine exercises - Baduanjin — According to the four steps of the cross-theoretical model, the behavior stage (pre-intention stage, intention stage, preparation stage, action stage and maintenance stage) and the family empowerment (clarify the problem, express the emotion, formulate the plan, implement the plan, and evaluate the effect). Combined with the characteristics of elderly patients after PCI, the cardiac rehabilitation management plan was designed focusing on the timing of cardiac rehabilitation, the way of health guidance, safety and compliance management.
  Other Names: Cross-theoretical model; Family empowerment
  Arms: Test group A; Test group B; Test group C

SUMMARY:
This study explores the effect of Internet based improved Baduanjin combined cross-theoretical model in family empowering cardiac rehabilitation for elderly patients with coronary heart disease after PCI, provides a scientific and reasonable case management plan for the rehabilitation of patients with coronary heart disease, and provides a reference for the development of scientific and refined cardiac rehabilitation case management suitable for elderly patients with PCI.

DETAILED DESCRIPTION:
In this study, a total of 120 elderly patients with coronary heart disease who underwent PCI in our hospital from July 2024 to July 2025 were selected, and an improved Baduanjin combined cross-theoretical model based on the Internet was applied to empower family cardiac rehabilitation management. The effect of this method on cardiac rehabilitation of elderly patients with coronary heart disease after PCI operation was evaluated by four indexes: cardiac function index, quality of life, medication compliance and satisfaction degree, and scientific guidance was provided for clinical cardiac rehabilitation practice.

ELIGIBILITY:
Inclusion Criteria:

* (1) All met the diagnostic criteria for coronary heart disease;
* (2) PCI was performed for the first time with clear indications of PCI surgery;
* (3) Postoperative condition was stable;
* (4) NYHA cardiac function grade I-II;
* (5) Age 60 ~75 years old;
* (6) Patients and their family members gave informed consent to this study and signed informed consent, which met the ethical standards of human trials and was approved by the ethics committee of the hospital.

Exclusion Criteria:

* (1) Uncontrolled arrhythmias combined with hemodynamic abnormalities.
* (2) COPD, pulmonary embolism, deep vein thrombosis, stroke and other factors affecting motor function.
* (3) Physical disability affecting safety and full participation in the experiment.
* (4) myocarditis, cardiomyopathy, liver and kidney insufficiency.
* (5) Aphasia, hearing impairment and other conditions affecting normal doctor-patient communication.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
left ventricular Ejection fraction (LVEF) | base line and 6 months after intervention
  Left ventricular ejection fraction (LVEF) was measured by echocardiography, and cardiac function was evaluated by the New York College of Cardiology (NYHA) grading standard. The detecting instrument is full digital color Doppler ultrasonic diagnosis instrument.

SECONDARY OUTCOMES:
Quality of life of patients after PCI | base line and 6 months after intervention
  Seattle Angina Pectoris Scale was used to evaluate the quality of life of patients after PCI.
Medication compliance | base line and 6 months after intervention
  The Questionnaire of Medication Compliance was adopted, including four questions, and each question was scored in four sections ranging from 1 to 4 points. The lowest score for each item was 1 point and the highest score was 4 points, that is, it could not be done at all =1, it could be done occasionally =2, it could be done basically =3, and it could be done completely =4. The score ranges from 0 to 16 points, and the higher the score, the better the patient's medication compliance. In this study, the reliability Cronbacha coefficient of the questionnaire was 0.875, and the content validity (CVI) value was 0.945.
The evaluation results of patient satisfaction at 6 months after intervention were compared between the groups | base line and 6 months after intervention
  the satisfaction was calculated by the unified survey of inpatient discharge satisfaction in our hospital, with a total score of 100, satisfaction > 90 points, unsatisfactory ≤90 points.

CONTACTS AND LOCATIONS:
Overall Officials: Shanshan Si, BA, Principal Investigator — 4th Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No